CLINICAL TRIAL: NCT05283330
Title: A Phase 1 Open-Label, First-in-human, Dose Escalation and Expansion Study to Determine the Safety, Tolerability, Dosimetry, Pharmacokinetics, and Preliminary Efficacy of 212Pb-DOTAM-GRPR1 in Adult Participants With Recurrent or Metastatic GRPR-expressing Tumors
Brief Title: Safety and Tolerability of ²¹²Pb-DOTAM-GRPR1 in Adult Subjects With Recurrent or Metastatic GRPR-expressing Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Orano Med LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OM-GRPR1-02
Record Dates: First submitted 2022-02-13; First posted 2022-03-16 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Cervical Cancer; Breast Cancer; Colon Cancer; NSCLC; mCRPC (Metastatic Castration-resistant Prostate Cancer); Glioblastoma; Nonsmall Cell Lung Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Breast Neoplasms; Colonic Neoplasms; Glioblastoma; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ²¹²Pb-DOTAM-GRPR1 (Experimental): In the dose escalation portion, a classic 3+3 design will be utilized for the SAD cohorts and a Boin design for the MAD cohorts. Doses will be increased by approximately 30% in subsequent cohorts. The maximum total dose that may be administered to a subject per cycle is 5.5 mCi +/- 10%.
  Interventions: Drug: ²¹²Pb-DOTAM-GRPR1

INTERVENTIONS:
Drug: ²¹²Pb-DOTAM-GRPR1 — ²¹²Pb-DOTAM-GRPR1 is a radioimmunoconjugate comprised of ²¹²Pb, the metal chelator DOTAM (1,4,7,10-Tetrakis(carbamoylmethyl)-1,4,7,10- tetraazacyclododecane) and a GRPR-targeted antagonist.

SUMMARY:
A Phase 1 Open-Label, First-in-human, Dose Escalation and Expansion Study to Determine the Safety, Tolerability, Dosimetry, Pharmacokinetics, and Preliminary Efficacy of 212Pb-DOTAM-GRPR1 in Adult Participants with Recurrent or Metastatic GRPR-expressing Tumors

DETAILED DESCRIPTION:
In this open-label, dose escalation and dose expansion single ascending dose (SAD) and multiple ascending dose (MAD) phase 1 study, participants with recurrent or metastatic histologically confirmed GRPR-expressing tumors will be enrolled. In the dose escalation portion, a classic 3+3 design will be utilized for the SAD cohorts and a BOIN design for the MAD cohorts. Dose escalation may proceed until the recommended MAD dose is determined. Up to six (2 SAD and 4 MAD) cohorts are expected to be enrolled. Participants will be treated with up to four cycles administered every 4 or 6 weeks. Once the recommended MAD dose is determined, the expansion cohorts of the study will commence. A dosimetry sub study will also be conducted in participants part of the dose escalation.

ELIGIBILITY:
1. Adult participants (age ≥ 18 years old) with any of the following advanced or metastatic solid tumors (documented history of histologically confirmed diagnosis):

   1. Metastatic castration-resistant prostate cancer (mCRPC) including neuroendocrine prostate cancer (NEPC) (enrolled only in SAD and MAD Q6W)
   2. HR+/HER2- breast cancer (estrogen receptor/ER expression >10% of tumor cell nuclei stain, regardless of progesterone receptor/PgR expression); HER2-negative including HER2-low (as per relevant ASCO/CAP guidelines)
   3. Colorectal cancer
   4. Cervical cancer
   5. Non-small-cell lung cancer (NSCLC)
   6. Recurrent glioblastoma (only enrolled in MAD Q4W cohorts) with evidence of recurrent disease (RD) demonstrated by disease progression using modified Response Assessment in Neuro-Oncology (RANO 2.0) criteria. Note: If surgery is performed for GBM recurrence, pre-surgery MRI will be used for confirmation of RD and residual and measurable disease post-surgery is not required but surgery must have confirmed the recurrence diagnosis by MRI.
2. Capable of giving signed informed consent
3. All participants must have progressed on at least 2 prior systemic therapies, except for recurrent GB
4. For participants with mCRPC: Prior orchiectomy and/or ongoing androgen deprivation therapy and a castrate level of serum testosterone (<50 ng/dL or <1.7 nmol/L)
5. Presence of at least 1 measurable lesion per RECIST 1.1 as assessed by the Investigator (not applicable for GBM). At least 1 identified measurable lesion must show GRPR uptake in 203Pb-DOTAM-GRPR1 SPECT/CT (uptake greater than that of the background) as assessed by the Investigator.
6. For participants with prostate cancer that do not have measurable soft tissue disease, 203Pb-DOTAM-GRPR1 uptake in bone lesions > uptake in background is acceptable for eligibility.
7. Eastern Cooperative Oncology Group (ECOG) status 0-1. Participants with ECOG status of 2 may be approved on a case-by-case basis in discussion with the Sponsor.
8. Adequate bone marrow, hepatic, and renal function, as assessed by the following laboratory requirements:

   1. White blood cell (WBC) ≥3000/ mm3 (≥ 3 x 109/L)
   2. Absolute neutrophil count (ANC) ≥1500/mm3 (≥1.5 x 109/L)
   3. Platelets ≥100,000/mm3 (≥ 100 x 109/L)
   4. Hemoglobin (Hb) ≥9.0 g/dL
   5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3x upper limit of normal (ULN) or ≤ 5 x ULN in the presence of liver metastases
   6. Total bilirubin: ≤1.5 x ULN, except if documented history of Gilbert's disease who are eligible if total bilirubin ≤ 3 x ULN
   7. Adequate renal function defined by creatinine clearance (CLCR) ≥ 60 mL/min calculated as follows: CLCR = eGFR in ml/min/1.73 m2 calculated by the Modified Diet in Renal Disease (MDRD) x participant body surface area (BSA) in m2 ÷ 1.73
   8. Serum amylase and/or lipase ≤1.5 x ULN
9. For women of childbearing potential (WOCBP) and men with partners of childbearing potential: be willing to use highly effective methods of contraception or sexual abstinence, if part of participant's lifestyle, throughout the study and for 7 months for WOCBP, 4 months for men after the last [212Pb]Pb-DOTAM-GRPR1 administration or for 10 days following [203Pb]Pb-DOTAM-GRPR1 administration and participant is not proceeding to 212Pb-DOTAM-GRPR1 treatment, as outlined in protocol.

   Participants with Recurrent Glioblastoma:
10. Having first or second glioblastoma recurrence, after standard therapy that includes prior radiation therapy (RT) and at least 12 weeks from completion of RT prior to first administration of 212Pb-DOTAM-GRPR1. In case surgery has been performed for GBM recurrence, the surgery has to be completed at least 4 weeks prior to 212Pb-DOTAM-GRPR1 treatment start, with post-surgery recovery without any complications related to surgical procedure.
11. Presence of 203Pb-DOTAM-GRPR1 uptake by SPECT/CT scan in the tumor lesion(s).
12. Presence of Gadolinium enhancement in the MRI in the tumor lesion(s) shown at the time of diagnosis of tumor recurrence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-12-22 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2032-05 (Estimated)

PRIMARY OUTCOMES:
To determine the Recommended Phase 2 Dose (RP2D) of ²¹²Pb-DOTAM-GRPR1 | 14 months
  Incidence of DLTs.

SECONDARY OUTCOMES:
To assess the safety and tolerability of 212Pb-DOTAM-GRPR1. | 24 months
  Measured as Incidence and severity of TEAEs and TESAEs.
To assess the safety and tolerability of 203Pb-DOTAM-GRPR1. | 24 months
  Measured as Incidence and severity of TEAEs and TESAEs.
To assess PK of ²¹²Pb-DOTAM-GRPR1 | 24 months
  212Pb-DOTAM-GRPR1 radioactivity concentration as a function of time in whole blood, plasma and urine
To evaluate the preliminary antitumor activity of 212Pb-DOTAM-GRPR1. | 24 months
  ORR by RECIST1.1, DOR, PFS by Investigator assessment and OS.
To evaluate the preliminary antitumor activity of 212Pb-DOTAM-GRPR1 | 24 months
  For participants with mCRPC, by Investigator assessment of ORR which is defined as a proportion of participants having a 'best overall response' (BOR) assessment of Complete Response (CR) or Partial Response (PR) as per PCWG3 guidelines.
To evaluate the preliminary antitumor activity of 212Pb-DOTAM-GRPR1 | 24 months
  For participants with mCRPC, by Investigator assessment of DOR which is defined as the time from the first documented objective response of PR or CR by PCWG3, whichever occurs earlier, to disease progression or death.
To evaluate the preliminary antitumor activity of 212Pb-DOTAM-GRPR1 | 24 months
  For participants with mCRPC, by Investigator assessment of PFS which is defined as the time from the start of study intervention to the date of first observed disease progression (Investigator's radiological assessment), clinical disease progression (Investigator's assessment) or death due to any cause as per PCWG3 guidelines.
To evaluate the preliminary antitumor activity of 212Pb-DOTAM-GRPR1 | 24 months
  For participants with mCRPC, as Overall Survival (OS) is defined as the time from the date of the start of study intervention to the date of death due to any cause.
To evaluate the preliminary antitumor activity of 212-PbDOTAM-GRPR1. | 24 Months
  For participants with recurrent GBM, by Investigator assessment of ORR which is defined as a proportion of participants having a 'best overall response' (BOR) assessment of Complete Response (CR) or Partial Response (PR) as per RANO 2.0 criteria.
To evaluate the preliminary antitumor activity of 212Pb-DOTAM-GRPR1. | 24 months
  For participants with recurrent GBM, by Investigator assessment of DOR defined as the time from the first documented objective response of PR or CR by RANO v 2.0, whichever occurs earlier, to disease progression or death
To evaluate the preliminary antitumor activity of 212Pb-DOTAM-GRPR1. | 24 months
  For participants with recurrent GBM, Investigator assessment of PFS defined as the time from the start of study intervention to the date of first observed disease progression (Investigator's radiological assessment), clinical disease progression (Investigator's assessment) or death due to any cause as per RANO 2.0 criteria.
To evaluate the preliminary antitumor activity of 212Pb-DOTAM-GRPR1. | 24 months
  For participants with recurrent GBM, Overall Survival (OS) is defined as the time from the date of the start of study intervention to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Northwestern University Robert H Lurie Medical Research, Chicago, Illinois
  - UK Markey Cancer Center, Lexington, Kentucky
  - Advanced Molecular Imaging and Therapy, Glen Burnie, Maryland
  - XCancer Omaha / Urology Cancer Center, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Taunk NK, Escorcia FE, Lewis JS, Bodei L. Radiopharmaceuticals for Cancer Diagnosis and Therapy: New Targets, New Therapies-Alpha-Emitters, Novel Targets. Cancer J. 2024 May-Jun 01;30(3):218-223. doi: 10.1097/PPO.0000000000000720. PMID 38753757
- [Derived] Kunos CA, Fabian D, Napier D, Stonecypher MS, Duncan RM, Hurt J. Human gastrin- releasing peptide receptor expression in women with uterine cervix cancer. Front Oncol. 2023 Jan 25;13:1126426. doi: 10.3389/fonc.2023.1126426. eCollection 2023. PMID 36761980